CLINICAL TRIAL: NCT07086235
Title: Randomized Split-Mouth Clinical Trial on Remineralization Capacity and Patient Satisfaction of Self-Assembling Peptide With Fluoride Versus Tooth Protective Coating With Surface Pre-Reacted Glass on White Spot Lesions
Brief Title: Remineralization Capacity and Patient Satisfaction of Self-Assembling Peptide With Fluoride Versus Tooth Protective Coating With Surface Pre-Reacted Glass on White Spot Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nahda University (Other)
Responsible Party: Principal Investigator, Khaled Wagih Al-Saudi, Lecturer of Operative and Conservative Dentistry, Nahda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00A-2-25-4
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: White Spot Lesions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Curodont Repair Fluoride Plus (Experimental)
  Interventions: Drug: self-assembling peptide
- S-PRG Barrier Coat (Experimental)
  Interventions: Drug: S-PRG Barrier Coat

INTERVENTIONS:
Drug: self-assembling peptide — According to the instructions of the manufacturer, the lesion will be treated with etch solution (Super Etch, SDI Ltd, Bayswater, Victoria, Australia) for 30 seconds to open up the pores to the subsurface lesion and subsequently will be washed and dried. Curodont Repair Fluoride Plus brush will be rehydrated with 0.05 ml of sterile water and a single drop of the resulting solution will be immediately applied to the lesion surface. Moisture control will be ensured until the Curodont Repair Fluoride Plus solution will be no longer visible (approximately two minutes).
  Arms: Curodont Repair Fluoride Plus
Drug: S-PRG Barrier Coat — According to the instructions of the manufacturer, after mixing one drop of activator with base, a thin film coating will be applied to the WSL area then will be left undistributed for 3 seconds and finally will be light cured for 10 seconds using LED light-curing unit.
  Arms: S-PRG Barrier Coat

SUMMARY:
Cosmetics and esthetics are current trends of our society, as more and more patients are demanding for minimally invasive cosmetic enhancement without anesthesia, drilling and less expensive restorations. This technique may be considered as micro invasive treatment of smooth surface white spot lesions (WSL) and also one that allows for the recovery of natural tooth appearance. Dentists are frequently faced with the treatment of color aberrations of teeth, as WSL which is caused by demineralization of enamel, and labial white spots are frequently associated with fixed orthodontic treatment. Clinically, the appearance of the lesion is opaque white, due to the optical phenomenon caused by mineral loss and the difference in the refractive index of water and air that fill the spaces formed in the enamel. The milky color of WSL impairs dramatically the esthetic appearance thus reducing satisfaction of orthodontic therapy, making their treatment become nowadays mandatory. Regarding the diagnosis, it is essential that the dentist does not lose the ability to detect a carious lesion or a WSL through visual or photographic examination, as is the most conventional way. However, other forms of diagnosis have emerged, such as fluorescence devices, as well as microradiography and microcomputed tomography to facilitate and accelerate the diagnostic process.

Conventionally, topical fluoride application has been used to manage WSLs in which the structure of the tooth is altered due to fluorapatite, thus becoming more resistant to caries. However, this approach has the disadvantage of depending on patient compliance and its results can be disappointing when solely used in high-risk patients. A recent biomimetic material has been introduced to dental market, namely, Curodont Repair Fluoride Plus, which is regarded as a possible substitute to fluoride to arrest WSL progression with the aim of filling the intercrystalline spaces for enamel subsurface lesions through a self-assembling peptide that builds a supramolecular three-dimensional, fibrous network in the acidic environment attracts calcium phosphate from saliva and produced de novo hydroxyapatite crystals surrounding the matrix with containing fluoride which have synergistic effect and enhance faster remineralization in management of WSLs. Another recent generation of patented bioactive smart remineralizing material, S-PRG Barrier Coat has been launched to remineralize WSLs where S-PRG pretreated fluoro-boro-aluminosilicate glass with polyacrylic acid and water to recharge and release fluoride. Additionally, releasing more types of ions this aid in biofilm suppression, decrease adhesion of bacteria, buffering capacity of acids, and enhances remineralization. The aim of this study is to compare the remineralization capacity and patient satisfaction of self-assembling peptide with fluoride versus tooth protective coating with surface pre-reacted glass on white spot lesions.

ELIGIBILITY:
Inclusion Criteria:

- No systemic diseases. 2- He/ she has at least two teeth with white spot lesion due to orthodontic therapy.

3- Between the ages of 21 and 25 years of age.

Exclusion criteria:

1. Presence of enamel hypoplasia or dental fluorosis.
2. Presence of tetracycline pigmentation.
3. Periodontal pocketing of 3 mm or greater.
4. Presencia de cavidades cariosas.
5. Allergy to fluoride.
6. Subjects who have evidence of reduced salivary flow or significant tooth wear.

Ages: 21 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2025-02-16 (Actual); Primary Completion 2025-08-16 (Actual); Study Completion 2025-08-16 (Actual)

PRIMARY OUTCOMES:
Color change assessment | Base-line (before treatment), immediately after treatment, 1-month, 3-month, and 6-months.
  Spectrophotometric color measurements will be performed using Vita Easy Shade (VITA Zahnfabrik, Germany). Only the lightness difference (ΔL*) value between baseline and after treatment will be recorded in this study.

SECONDARY OUTCOMES:
Depth of White Spot Lesions | Base-line (before treatment), immediately after treatment, 1-month, 3-months, and 6-months.
  The depth of all lesions from all subjects will be assessed using DIAGNOdent (KaVo, Germany), which relies on measuring the amount of fluorescence released by organic substances in dental tissues when stimulated by a 655 nm laser diode.

OTHER OUTCOMES:
Patient satisfaction | Base-line (before treatment), immediately after treatment, 1-month, 3-months, and 6-months.
  Patient satisfaction will be assessed using the visual Analog Scale Score (VAS). The VAS is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points. A 10 cm line with the anchor words "no sensitivity" at one end and "intolerable sensitivity" at the other end.

CONTACTS AND LOCATIONS:
Locations (1):
- Nahda University, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No